CLINICAL TRIAL: NCT06011239
Title: Family Teams: A Study to Promote Team Collaboration in Family Medicine Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Katherine Gold, Associate Professor of Family Medicine and of Obstetrics and Gynecology, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00239209
Record Dates: First submitted 2023-08-18; First posted 2023-08-25 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Patient Care Team; Psychological Well-Being; Occupational Burnout
Keywords: family medicine; team function; burnout; compassion
MeSH Terms: conditions — Psychological Well-Being; Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: The study will recruit all staff except the clinic managers at each of five family medicine clinics within our academic family medicine department.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Survey participants (Experimental): All participants in the study will be in a single arm, divided by clinic.
  Interventions: Behavioral: Team-building processes
- Clinic Staff (No Intervention): "Project champions" at each clinic who are helping to implement the project.

INTERVENTIONS:
Behavioral: Team-building processes — All staff in one of the four role groups (medical assistants (MAs); clerical/administrative staff; nursing staff; and physicians/nurse practitioners/physician assistants) will be sent an anonymous survey. The survey will ask staff to consider what help participants wish to ask for and what help participants can offer to staff in the other three roles at times when people are busy or overwhelmed. These ideas will be combined into a typed "idea list" for each role and then staff in clinics will discuss. Once these are finalized the clinics will implement these.
  At several points during the year, the study team will send out brief surveys. These surveys will collect the clinic and job role and ask participant to rate how much effort has been made in different ways, and if there are open-ended comments about what is or is not working. This information will be used to improve the intervention at each clinic.
  Arms: Survey participants

SUMMARY:
This project includes an intervention in five Michigan Medicine family medicine clinics which is designed to improve staff collaboration across different job roles.

DETAILED DESCRIPTION:
The primary intervention asks staff to meet with others in the same role and to consider the following questions:

* The Ask: When staff are busy or overwhelmed by work, what tasks can others do (people in each of these groups) to help make your job better or easier?
* The Offer: When people in other groups are busy or overwhelmed, what tasks can your group do to help make staff jobs better or easier?

After this information is collected, at an in-person meeting of all staff and faculty, the study team will divide everyone into groups by clinic and then by the four roles. The study team will hand out the idea list and ask participants to review the list, discuss whether there are new or additional ideas which should be added, and then prioritize staffs top five "asks" and top five "offers" for staff role.

Negotiation of asks/offers: The study team will hold 1-4 subsequent brief meetings at each clinic where staff are again sub-divided into four groups by role. Each group will review the asks from people in other roles and decide whether these are actions that staff can help with or whether there are barriers. The clinic champions will work with the groups to address barriers (which could include lack of information, lack of training, disagreements about need, etc). The ultimate goal will be for groups to come to consensus agreement on at least three ways staff can assist people in other roles. In some clinics this may be straightforward and require just one meeting. In other clinics, it may take several meetings.

Implementation: Once the asks and offers are finalized, it will be up to the physician champions to help promote these agreements at the clinic, follow up with staff and with the nursing, medical assistants, and clerical champions to ensure that people are following thru with commitments to help, and trouble shoot problems that come up.

Coordination with Leadership: a department leader will serve as the liaison between the clinic champions and members of leadership that oversee clinical functions. This leader meets regularly with these leadership groups and will help troubleshoot challenges to implementing the asks and offers which need higher-level approval or input.

Ongoing process improvement: Over time, the study team will send up to four brief, anonymous surveys to all staff asking whether the staff are indeed doing the things that staff committed to do and whether other role groups are following thru on the commitments. This provides an opportunity for people to identify and report problems. This data will be anonymously fed back to the physician champion that is tasked to troubleshoot and address the problems identified, working with the liaison as appropriate. This will likely require continuous process improvement and revisiting to ensure success.

Evaluation: The study team proposes to measure burnout and team centeredness using anonymous on-line surveys.

Brief surveys: At several points during the year, the investigators will send out brief surveys. These ask for the clinic and job role and then ask participant to rate how much effort they have made to help others, how much effort others have made to help them, and if there are open-ended comment about what is or is not working. This information will be used to improve the intervention at each clinic.

Qualitative interviews regarding clinic culture will also be conducted with the project champions at each clinic who are helping to implement the project.

This study is Institutional review board (IRB) exempt and will have a waiver of documentation of informed consent with survey completion representing consent.

ELIGIBILITY:
Inclusion Criteria:

* Staff in the roles of medical assistant, nurse, clerical staff, or clinician (physician, nurse practitioner, and physician assistant)
* Must work in one of five family medicine clinics at the University of Michigan.

Exclusion Criteria:

* administrative clinic director at each site (managerial)
* Staff outside of the above roles such as a dietician, social worker, pharmacist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Team Development measure | Months 0, 12, 18
  The Team Development Measure is a 31-item questionnaire designed to the domains of communication, roles and goals, cohesion, and team primacy. Each question has four response options (strongly disagree, disagree, agree, strongly agree). Summary scores are transformed to a 0-100 scale to provide a score of team functioning and cohesiveness with a higher score indicating a better-functioning team. This measure has been validated in primary care settings and has strong psychometric properties.
Team Compassion Behavior survey | Months 0, 12, 18
  The Team Compassion Behavior survey is a 6-question instrument adapted for teams from a longer individual compassion instrument. It is scored on a 5-point scale (almost never, seldom, sometimes, often, almost always) and summed for a total range of 6-30 point, with a higher score indicating more compassionate team behavior.
Burnout | Months 0, 12, 18
  The study team will use the first 10 questions of the Mini Z 3.0 (the 11th question is open-ended) to measure burnout across staff in all roles. It has just minor changes from the earlier MiniZ versions and has good performance with two subscales for supportive work environment and electronic medical record (EMR) stress. Each question has a 5-scale response option. Subscale 1 (supportive work environment) sums the responses to questions 1-7 and has a range of 7-35 with a score of 28 or higher indicating a highly supportive workplace. Subscale 2 (EMR stress) sums responses to questions 8-10 and has a range of 3-15 with a score of 12 or higher indicating a workplace with manageable EMR stress.
Satisfaction with Intervention | Months 0, 12, 18
  There are several open-ended questions to assess what is working well with the project, what could be improved, and any other comments about the intervention. There is also a question asking how participants feel about the project (5-point scale ranging from extremely negative to extremely positive).
Participation Effort | Months 0, 12, 18
  This survey asks to report how much effort participants have made to help other groups in clinic and how much effort each of the other groups have made to help them. These questions have a 5-point scale (none at all, a little, a moderate amount, a lot, a great deal). These surveys also ask two open ended questions: problems with the intervention and what is not working in clinic with respect to the project and what is working well. This data will help the study team do continuous quality improvement within the clinics to ensure that the agreed-upon help is actually occurring.

OTHER OUTCOMES:
Clinic Culture | 1 month
  Project champions (clinic staff who are helping implement the project) will participate in interviews from which qualitative data about clinic culture will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Gold, MD, Principal Investigator — University of Michigan
Locations (5):
- United States (5):
  - University of Michigan-Domino Farms, Ann Arbor, Michigan
  - University of Michigan- Briarwood, Ann Arbor, Michigan
  - Uniiversity of Michigan- Chelsea, Chelsea, Michigan
  - University of Michigan-Dexter, Dexter, Michigan
  - University of Michigan-Ypsilanti, Ypsilanti, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stock R, Mahoney E, Carney PA. Measuring team development in clinical care settings. Fam Med. 2013 Nov-Dec;45(10):691-700. PMID 24347186
- [Background] Wee EXM, Fehr R. Compassion during difficult times: Team compassion behavior, suffering, supervisory dependence, and employee voice during COVID-19. J Appl Psychol. 2021 Dec;106(12):1805-1820. doi: 10.1037/apl0001001. PMID 34968091
- [Background] Pommier E, Neff KD, Toth-Kiraly I. The Development and Validation of the Compassion Scale. Assessment. 2020 Jan;27(1):21-39. doi: 10.1177/1073191119874108. Epub 2019 Sep 13. PMID 31516024
- [Background] Linzer M, McLoughlin C, Poplau S, Goelz E, Brown R, Sinsky C; AMA-Hennepin Health System (HHS) burnout reduction writing team. The Mini Z Worklife and Burnout Reduction Instrument: Psychometrics and Clinical Implications. J Gen Intern Med. 2022 Aug;37(11):2876-2878. doi: 10.1007/s11606-021-07278-3. Epub 2022 Jan 19. No abstract available. PMID 35048290